CLINICAL TRIAL: NCT00911170
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study of Pegfilgrastim Admininstered to Subjects With Newly Diagnosed, Locally-advanced or Metastatic Colorectal Cancer Treated With Bevacizumab & Either 5-fluorouracil, Oxaliplatin, Leucovorin (FOLFOX) or 5-fluorouracil, Irinotecan, Leucovorin (FOLFIRI)
Brief Title: PAVES: Pegfilgrastim Anti-vascular Endothelial Growth Factor (VEGF) Evaluation Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20080259
Record Dates: First submitted 2009-05-21; First posted 2009-06-01 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Cancer; Colon Cancer; Colorectal Cancer; Fever; Locally Advanced; Metastatic Colorectal Cancer; Neutropenia; Rectal Cancer
Keywords: adenocarcinoma of the colon or rectum; febrile neutropenia; Bevacizumab; Avastin; 5-fluorouracil, Oxaliplatin, Leucovorin (FOLFOX); 5-fluorouracil, Irinotecan, Leucovorin (FOLFIRI)
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Colorectal Neoplasms; Fever; Neutropenia; Rectal Neoplasms; Febrile Neutropenia | interventions — pegfilgrastim; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received standard chemotherapy (FOLFOX or FOLFIRI) on Days 1-2, and bevacizumab 5 mg/kg intravenous (IV) infusion on Day 1 of each 14-day cycle plus placebo subcutaneous injection once per cycle, for a maximum of 4 cycles, 24 hours after chemotherapy (Day 4).
  Interventions: Drug: Placebo; Biological: Bevacizumab; Drug: Standard Chemotherapy
- Pegfilgrastim (Placebo Comparator): Participants received standard chemotherapy (FOLFOX or FOLFIRI) on Days 1-2 and bevacizumab 5 mg/kg intravenous (IV) infusion on Day 1 of each 14-day cycle plus pegfilgrastim 6 mg administered as a single subcutaneous injection once per cycle, for a maximum of 4 cycles, 24 hours after chemotherapy (Day 4).
  Interventions: Drug: Pegfilgrastim; Biological: Bevacizumab; Drug: Standard Chemotherapy

INTERVENTIONS:
Drug: Pegfilgrastim — Administered as a single 6 mg subcutaneous injection using a pre-filled syringe. There will be no dosage adjustments for investigational product.
  Other Names: Neulasta®
  Arms: Pegfilgrastim
Drug: Placebo — Administered as a single subcutaneous injection using a pre-filled syringe.
  Arms: Placebo
Biological: Bevacizumab — 5 mg/kg by intravenous (IV) infusion on day 1 of each 14-day cycle.
  Other Names: Avastin®
Drug: Standard Chemotherapy — Each participant received one of the following chemotherapy regimens at the discretion of treating physician:
  FOLFOX: Oxaliplatin, leucovorin, and 5-fluorouracil; FOLFIRI: Irinotecan, leucovorin and 5-flurouracil.

SUMMARY:
This is a phase 3, randomized, double-blind, placebo-controlled multi-center study evaluating the efficacy of pegfilgrastim to reduce the incidence of febrile neutropenia (FN) in patients with newly diagnosed, locally-advanced or metastatic colorectal cancer receiving first-line treatment with bevacizumab and either 5-fluorouracil, Oxaliplatin, Leucovorin (FOLFOX) or 5-fluorouracil, Irinotecan, Leucovorin (FOLFIRI).

This study will also investigate the effect of adding pegfilgrastim to bevacizumab and either FOLFOX or FOLFIRI by evaluating overall survival, progression-free survival, and overall response rate in each arm at regular intervals over a maximum of 60 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

Disease-related:

* Histologically or cytologically-confirmed adenocarcinoma of the colon or rectum
* Locally-advanced or metastatic disease by radiographic evaluation
* Measurable disease
* Has not previously received chemotherapy for locally-advanced or metastatic colorectal cancer. Patient may have received adjuvant therapy for primary colorectal cancer provided that at least 6 months have elapsed from the time the adjuvant therapy was concluded and recurrent/metastatic disease was documented.
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2

Demographic:

- Age of 18 years or over

Laboratory:

Adequate organ and marrow function as defined below:

* Absolute neutrophil count at least 1.5 x 10^9/L
* Platelet count at least 100 x 10^9/L
* Bilirubin ≤ 1.5 times upper limit of normal
* Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x upper limit of normal or Aspartate aminotransferase and alanine aminotransferase ≤ 5.0 x upper limit of normal if attributable to liver metastasis
* An in-range international normalized ratio (INR) (in-range is usually defined as between 2 and 3) for patients on a stable dose of oral anticoagulant or stable dose of low molecular weight heparin
* Has no active bleeding or pathological condition that carries high risk of bleeding (eg, tumor involving major vessels or known varices). If a suspicion of bleeding diathesis exists, a bleeding time should be performed
* Creatinine ≤ 1.5 times upper limit of normal

General:

* Written informed consent obtained
* Afebrile on day 1 of cycle 1
* Must be able and willing to comply with study and/or follow-up procedures

Exclusion Criteria:

Disease-Related:

* Known brain metastases
* History of another primary malignancy less than/equal to 5 years prior to randomization, with the exception of non-melanoma skin cancer, carcinoma in situ of uterine cervix, and prostatic intraepithelial neoplasia without evidence of prostate cancer
* Prior major surgical procedure less than 28 days prior to day 1 of cycle 1 chemotherapy dosing; anticipated need for major surgical procedure during the 4 cycle treatment period of the study
* Fine needle aspirations or core biopsies within 7 days prior to day 1 of cycle 1 chemotherapy dosing
* Serious nonhealing wound, ulcer, or bone fracture, or history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to day 1 of cycle 1
* Uncontrolled high blood pressure, history of labile hypertension, uncontrolled congestive heart failure, unstable angina within the past 3 months, myocardial infarction or history of stroke within the past 12 months, unstable symptomatic arrhythmia requiring medication, or clinically significant peripheral vascular disease
* History of clinically significant bleeding within 6 months prior to randomization
* History of arterial or venous thromboembolism within 6 months prior to randomization
* History of other disease including uncontrolled diabetes, serious active or uncontrolled infection, metabolic dysfunction; physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of the prescribed therapy or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications

Laboratory:

- Proteinuria > 1+, or total quantitative protein > 500 mg protein/day as determined by 24-hr urine collection

Medications:

* Prior radiotherapy unless treatment was limited to the target lesion and only 1 measurable lesion was treated. Progression of the irradiated lesion must be demonstrated. Patients may not have received prior radiotherapy to greater than 25% of bone marrow. Radiation must have concluded ≥ 4 weeks prior to enrollment. Prior radio-sensitizing chemoradiation will be allowed as long as it was concluded ≥ 4 weeks prior to enrollment.
* Radiotherapy to non-target lesions for pain control will be allowed
* Prior bevacizumab use or other agents targeting VEGF
* Concurrent use of other biological agents
* Use of systemic anti-infectives for active infection, during the 3 calendar days before starting study chemotherapy and bevacizumab or planned during the study treatment period

General:

* Current, recent (within 4 weeks of the first infusion of this study), or planned participation (during the study treatment period) in an experimental therapeutics study other than this protocol
* Female participants who are pregnant or lactating or men and women of reproductive potential not willing to employ an effective method of birth control during treatment and for 20 weeks for women, and 30 weeks for men after discontinuing study treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab, irinotecan, 5-fluorouracil (5-FU), oxaliplatin, or leucovorin, including known sensitivity to E. Coli derived products (eg, Filgrastim, HUMULIN insulin, L-asparaginase)
* Known dihydropyrimidine dehydrogenase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 847 (Actual)
Dates: Start 2009-11-03 (Actual); Primary Completion 2012-09-17 (Actual); Study Completion 2015-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (142):
- United States (69):
  - Research Site, Muscle Shoals, Alabama
  - Research Site, Jonesboro, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Modesto, California
  - Research Site, San Diego, California
  - Research Site, Greenwich, Connecticut
  - Research Site, Dover, Delaware
  - Research Site, Gainesville, Florida
  - Research Site, Loxahatchee Groves, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Gurnee, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Quincy, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, New Albany, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Council Bluffs, Iowa
  - Research Site, Sioux City, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, Hutchinson, Kansas
  - Research Site, Hazard, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Bethesda, Maryland
  - Research Site, Cumberland, Maryland
  - Research Site, Randallstown, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Jefferson City, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Grand Island, Nebraska
  - Research Site, Kearney, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Little Silver, New Jersey
  - Research Site, Somerville, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Lake Success, New York
  - Research Site, Nyack, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Massillon, Ohio
  - Research Site, Middletown, Ohio
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Reading, Pennsylvania
  - Research Site, Upland, Pennsylvania
  - Research Site, West Reading, Pennsylvania
  - Research Site, Willow Grove, Pennsylvania
  - Research Site, Hilton Head Island, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Bryan, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Abingdon, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Kennewick, Washington
  - Research Site, Spokane, Washington
- Australia (5):
  - Research Site, Hobart, Tasmania
  - Research Site, Ballarat, Victoria
  - Research Site, Coburg, Victoria
  - Research Site, Footscray, Victoria
  - Research Site, Frankston, Victoria
- Belgium (3):
  - Research Site, Aalst
  - Research Site, Roeselare
  - Research Site, Verviers
- Bulgaria (2):
  - Research Site, Sofia
  - Research Site, Varna
- Canada (8):
  - Research Site, Brampton, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, London, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
- Czechia (4):
  - Research Site, Hořovice
  - Research Site, Nová Ves pod Pleší
  - Research Site, Olomouc
  - Research Site, Znojmo
- France (5):
  - Research Site, Amiens
  - Research Site, Bordeaux
  - Research Site, Cahors
  - Research Site, Lille
  - Research Site, Rouen
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Szeged
  - Research Site, Szolnok
- Ireland (4):
  - Research Site, Cork
  - Research Site, Dublin
  - Research Site, Galway
  - Research Site, Waterford
- Italy (5):
  - Research Site, Benevento
  - Research Site, Palermo
  - Research Site, Roma (RM)
  - Research Site, Rozzano (MI)
  - Research Site, Taormina (ME)
- Latvia (2):
  - Research Site, Daugavpils
  - Research Site, Riga
- Mexico (3):
  - Research Site, San Luis Potosí City, San Luis P
  - Research Site, Colima
  - Research Site, Toluca
- Poland (5):
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Suwałki
  - Research Site, Warsaw
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Sibiu
- Russia (6):
  - Research Site, Chelyabinsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Yaroslavl
- Slovakia (4):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Rimavská Sobota
  - Research Site, Trnava
- Ukraine (6):
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Uzhhorod

REFERENCES:
- [Background] Pinter T, Klippel Z, Cesas A, Croitoru A, Decaestecker J, Gibbs P, Hotko Y, Jassem J, Kurteva G, Novotny J, O'Reilly S, Salek T, Reiner M, Morrow PK, Choi MR, Whittaker S, Blanke C. A Phase III, Randomized, Double-Blind, Placebo-Controlled Trial of Pegfilgrastim in Patients Receiving First-Line FOLFOX/Bevacizumab or FOLFIRI/Bevacizumab for Locally Advanced or Metastatic Colorectal Cancer: Final Results of the Pegfilgrastim and Anti-VEGF Evaluation Study (PAVES). Clin Colorectal Cancer. 2017 Jun;16(2):103-114.e3. doi: 10.1016/j.clcc.2016.08.008. Epub 2016 Sep 7. PMID 28038865
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled into the study on 03 November 2009 and the last participant on 03 January 2012.
Pre-assignment Details: This study included a a study treatment period (approximately 8 weeks), and a long-term follow-up period (up to 36 months after the last participant was enrolled).
Groups:
- Placebo: Participants received standard chemotherapy (FOLFOX or FOLFIRI) on Days 1-2, and bevacizumab 5 mg/kg intravenous (IV) infusion on Day 1 of each 14-day cycle, plus placebo subcutaneous injection once per cycle, for a maximum of 4 cycles, 24 hours after chemotherapy (Day 4). During the long-term follow-up period, further chemotherapy and/or biologic agents (for example, bevacizumab) were to continue at the discretion of the treating physician.
- Pegfilgrastim: Participants received standard chemotherapy (FOLFOX or FOLFIRI) on Days 1-2 and bevacizumab 5 mg/kg intravenous (IV) infusion on Day 1 of each 14-day cycle plus pegfilgrastim 6 mg administered as a single subcutaneous injection once per cycle, for a maximum of 4 cycles, 24 hours after chemotherapy (Day 4). During the long-term follow-up period, further chemotherapy and/or biologic agents (for example, bevacizumab) were to continue at the discretion of the treating physician.
Period: Treatment Period
Arm/Group | Placebo | Pegfilgrastim
Started | 424 | 423
Received Chemotherapy | 423 (Primary Analysis Set) | 422 (Primary Analysis Set)
Received Bevacizumab | 423 | 420
Received Investigational Product | 422 (Includes one participant who received pegfilgrastim in error.) | 419
Completed | 397 (Completed 4 cycles of treatment including chemotherapy, bevacizumab and investigational product.) | 386 (Completed 4 cycles of treatment including chemotherapy, bevacizumab and investigational product.)
Not Completed | 27 | 37
Not completed — Randomized in error | 1 | 1
Not completed — Ineligibility determined | 1 | 3
Not completed — Protocol deviation | 1 | 2
Not completed — Adverse Event | 9 | 10
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Disease progression | 0 | 2
Not completed — Physician Decision | 5 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 6 | 9
Period: Long Term Follow-Up
Arm/Group | Placebo | Pegfilgrastim
Started | 423 (Participants who received treatment in the Treatment Period) | 422 (Participants who received treatment in the Treatment Period)
Completed | 0 (As of the data cut-off date of 8 June 2012) | 0 (As of the data cut-off date of 8 June 2012)
Not Completed | 423 | 422
Not completed — Continuing in study | 274 | 269
Not completed — Withdrawal by Subject | 20 | 21
Not completed — Physician Decision | 5 | 4
Not completed — Lost to Follow-up | 8 | 7
Not completed — Death | 116 | 121

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received standard chemotherapy (FOLFOX or FOLFIRI) on Days 1-2, plus bevacizumab 5 mg/kg intravenous (IV) infusion on Day 1 of each 14-day cycle plus placebo subcutaneous injection once per cycle, for a maximum of 4 cycles, 24 hours after chemotherapy (Day 4).
- Total: Total of all reporting groups
Arm/Group | Placebo | Pegfilgrastim | Total
Number analyzed (Participants) | 423 | 422 | 845
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.7) | 60.6 (10.4) | 60.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 174 | 333
  Male | 264 | 248 | 512
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 2 | 5
  Black or African American | 6 | 4 | 10
  Hispanic or Latino | 8 | 11 | 19
  Japanese | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  White | 404 | 402 | 806
Chemotherapy Regimen [Number; unit: participants]
  FOLFOX | 207 | 207 | 414
  FOLFIRI | 216 | 215 | 431
Region [Number; unit: participants] — North America (Canada and the US) and the Rest of World (Australia, Belgium, Bulgaria, Czech Republic, France, Hungary, Ireland, Italy, Latvia, Mexico, Poland, Romania, Russian Federation, Slovakia, and Ukraine)
  participants
    North America | 79 | 77 | 156
    Rest of World | 344 | 345 | 689
Disease Status [Number; unit: participants]
  Locally Advanced | 18 | 18 | 36
  Metastatic | 405 | 404 | 809
Primary Tumor Diagnosis [Number; unit: participants]
  Colon | 284 | 290 | 574
  Rectum | 139 | 132 | 271

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 3/4 Febrile Neutropenia Across the First 4 Cycles of Chemotherapy
Description: Grade 3/4 febrile neutropenia (FN) is defined as: • A temperature ≥ 38.0°C (≥ 100.4°F) and absolute neutrophil count (ANC) < 1.0 × 10^9/L, where ANC was measured the same day or within ± 1 calendar day of a temperature ≥ 38.0°C (≥ 100.4°F), or • An ANC < 1.0 × 10^9/L in combination with: - documented sepsis or infection, OR - neutropenia-related hospitalization where ANC was measured the same day or within ± 1 calendar day. Participants monitored their oral temperatures and maintained diaries to record their temperature twice per day: once in the morning and once in the evening, as well as whenever they suspect they had fever throughout the first 4 cycles of chemotherapy treatment.
Time Frame: Approximately 2 months duration (Daily for 4 cycles of treatment; 2 weeks per cycle)
Population: The primary analysis set which included all participants with a signed informed consent, and who were randomized and received at least 1 dose of protocol-specified study treatment (chemotherapy, bevacizumab, or investigational product).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Pegfilgrastim
Number analyzed (Participants) | 423 | 422
percentage of participants | 5.7 [3.7 to 8.3] | 2.4 [1.1 to 4.3]
Statistical Analysis 1: Comparison: Placebo vs Pegfilgrastim; The primary hypothesis was that the percentage of participants treated with study chemotherapy and bevacizumab who experience grade 3/4 febrile neutropenia (FN) would be lower in participants randomized to the pegfilgrastim arm compared to placebo arm. The study was designed to have at least 90% power at the 2-sided 0.05 significance level to detect a 6% difference in incidence of grade 3/4 FN from 9% to 3%, which is approximately a 66.7% relative reduction; Test type: Superiority or Other; p = 0.014, Cochran-Mantel-Haenszel; The p-value is adjusted for the randomization stratification factors (chemotherapy regimen, geographic region, disease stage); Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.19 to 0.86] — Odds ratio adjusted for the randomization stratification factors. An OR < 1.0 indicates a lower event rate for the pegfilgrastim arm relative to the placebo arm

2. Secondary Outcome: Overall Survival
Description: Median time from randomization to date of death caclulated using the Kaplan-Meier method. Participants were censored on the date of last contact (i.e., the date the participant was last known to be alive) if they were not known to have died.
Time Frame: From randomization to the data cut-off date of 8 June 2012. Median time on study was 11.6 months and the maximum was 27.6 months.
Population: Primary analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Pegfilgrastim
Number analyzed (Participants) | 423 | 422
months | 24.6 [21.3 to NA] — Could not be estimated due to the low number of events. | 21.8 [18.5 to 25.6]
Statistical Analysis 1: Comparison: Placebo vs Pegfilgrastim; Test type: Superiority or Other; p = 0.704, Log Rank; P-values based on the log-rank test statistic from the Kaplan-Meier survival analysis stratified by the 3 randomization factors; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.81 to 1.36] — Based on Cox proportional Hazard model stratified by chemotherapy regimen, region and disease status. A HR< 1.0 indicates a lower average event rate and a longer survival time for the pegfilgrastim arm relative to the placebo arm

3. Secondary Outcome: Progression Free Survival
Description: Time from randomization to date of radiological disease progression or death from any cause, whichever event occurs first, calculated using the Kaplan-Meier method. Participants without either event by the analysis data cutoff date were censored on the date of their last evaluable disease assessment. Disease progression based on the investigator's assessment of radiographic scans using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Clinical progression without radiological assessment was not be considered a disease progression in this analysis. Progression defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 2
Population: Primary analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Pegfilgrastim
Number analyzed (Participants) | 423 | 422
months | 10.1 [9.3 to 11.1] | 9.7 [9.2 to 10.8]
Statistical Analysis 1: Comparison: Placebo vs Pegfilgrastim; Test type: Superiority or Other; p = 0.552, Log Rank; P-values are based on the log-rank test statistic from the Kaplan-Meier survival analysis stratified by the 3 randomization factors; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.88 to 1.26] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Time to Progression
Description: Time from randomization to date of radiological disease progression calculated using the Kaplan-Meier method. Participants without progression were censored on the date of their last radiographic tumor assessment. Disease progression based on the investigator's assessment of scans using the RECIST v1.1. Clinical progression without radiological assessment was not considered a disease progression. Progression defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 2
Population: Primary analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Pegfilgrastim
Number analyzed (Participants) | 423 | 422
months | 11.1 [10.0 to 11.8] | 10.8 [9.5 to 11.3]
Statistical Analysis 1: Comparison: Placebo vs Pegfilgrastim; Test type: Superiority or Other; p = 0.502, Log Rank; [statistical method as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.88 to 1.29] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Percentage of Participants With an Objective Response
Description: The percentage of participants with a complete response (CR) or partial response (PR) defined by the RECIST v1.1 criteria at any time during the study. Response was be determined by the investigator's assessment of radiographic scans. CR: Disappearance of all non-nodal target lesions and the disappearance of all non-nodal non-target lesions, and no new lesions. All nodal lesions must have reduction of short axis to < 10 mm. PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters and no new lesions and/or unequivocal progression of existing non-target lesions, or, the disappearance of all non-nodal target lesions with persistence of one or more non-target lesion(s).
Time Frame: as for outcome 2
Population: Primary analysis set participants with measurable disease at Baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Pegfilgrastim
Number analyzed (Participants) | 420 | 420
percentage of participants | 56.7 [51.8 to 61.5] | 58.1 [53.2 to 62.9]
Statistical Analysis 1: Comparison: Placebo vs Pegfilgrastim; Test type: Superiority or Other; p = 0.683, Cochran-Mantel-Haenszel; The p-value is from the Cochran Mantel Haenszel (CMH) test adjusting for the randomization stratification factors; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.81 to 1.39] — Odds ratio (OR) adjusted for the randomization stratification factors. An OR > 1.0 indicates a higher event rate for the pegfilgrastim arm relative to the placebo arm

6. Secondary Outcome: Percentage of Participants With Grade 4 Febrile Neutropenia Across the First 4 Cycles of Chemotherapy
Description: Grade 4 febrile neutropenia (FN) is defined as:
  * A temperature ≥ 38.0ºC (≥ 100.4ºF) and absolute neutrophil count (ANC) < 0.5 × 10^9/L, where ANC is measured the same day or within +/- 1 calendar day of a temperature ≥ 38.0ºC (≥ 100.4ºF), or
  * An ANC <0.5 × 10^9/L in combination with:
    * Documented sepsis or infection, OR
    * Neutropenia-related hospitalization where ANC is measured the same day or within +/- 1 calendar day.
Time Frame: Approximately 2 months duration (Daily for 4 cycles of treatment; 2 weeks per cycle)
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Pegfilgrastim
Number analyzed (Participants) | 423 | 422
percentage of participants | 3.5 [2.0 to 5.8] | 2.4 [1.1 to 4.3]
Statistical Analysis 1: Comparison: Placebo vs Pegfilgrastim; Test type: Superiority or Other; p = 0.312, Cochran-Mantel-Haenszel; The p-value is from the Cochran Mantel Haenszel (CMH) test adjusting for the randomization stratification factors; Odds Ratio (OR) = 0.66, 95% CI [0.29 to 1.49] — Odds ratio (OR) adjusted for the randomization stratification factors. An OR < 1.0 indicates a lower event rate for the pegfilgrastim arm relative to the placebo arm

7. Secondary Outcome: Percentage of Participants With Grade 3/4 Neutropenia Across the First 4 Cycles of Chemotherapy
Description: Grade 3/4 severe neutropenia is defined as neutropenia with absolute neutrophil count (ANC) <1.0 x 10^9/L.
Time Frame: Approximately 2 months duration (Daily for 4 cycles of treatment; 2 weeks per cycle)
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Pegfilgrastim
Number analyzed (Participants) | 423 | 422
percentage of participants | 17.0 [13.6 to 20.9] | 3.6 [2.0 to 5.8]
Statistical Analysis 1: Comparison: Placebo vs Pegfilgrastim; Test type: Superiority or Other; p < .001, Cochran-Mantel-Haenszel; The p-value is from the Cochran Mantel Haenszel (CMH) test adjusting for the randomization stratification factors; Odds Ratio (OR) = 0.18, 95% CI [0.10 to 0.32] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Percentage of Participants With Grade 4 Neutropenia Across the First 4 Cycles of Chemotherapy
Description: Grade 4 severe neutropenia is defined as neutropenia with absolute neutrophil count (ANC) <0.5 x 10^9/L.
Time Frame: Approximately 2 months duration (Daily for 4 cycles of treatment; 2 weeks per cycle)
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Pegfilgrastim
Number analyzed (Participants) | 423 | 422
percentage of participants | 8.3 [5.8 to 11.3] | 2.4 [1.1 to 4.3]
Statistical Analysis 1: Comparison: Placebo vs Pegfilgrastim; Test type: Superiority or Other; p < .001, Cochran-Mantel-Haenszel; The p-value is from the Cochran Mantel Haenszel (CMH) test adjusting for the randomization stratification factors; Odds Ratio (OR) = 0.27, 95% CI 2-sided [0.13 to 0.56] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: A serious adverse event (SAE) is defined as an adverse event that - is fatal; - is life threatening (places the participant at immediate risk of death); - requires inpatient hospitalization or prolongation of existing hospitalization; - results in persistent or significant disability/incapacity; - is a congenital anomaly/birth defect; - other significant medical hazard. AEs were assessed for severity according to National Cancer Institute, Common Terminology Criteria for Adverse Events, Version 3.0, based on this general guideline: Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE; Grade 5 = Death related to AE.
Time Frame: Approximately 8 weeks (4 treatment cycles)
Population: Safety analysis set, defined as all participants in the Primary Analysis Set who received at least one dose of investigational product (IP; placebo or pegfilgrastim). One participant was randomized to the placebo arm but actually received pegfilgrastim and is included in the pegfilgrastim arm for the safety analyses.
Measure: Number; unit: participants
Arm/Group | Placebo | Pegfilgrastim
Number analyzed (Participants) | 421 | 420
participants
  Any adverse event | 355 | 344
  Worst Grade of > 2 | 254 | 240
  Worst Grade of > 3 | 119 | 115
  Worst Grade of > 4 | 45 | 31
  Serious adverse events | 55 | 68
  Severe adverse events | 103 | 106
  Life-threatening adverse events | 43 | 27
  Fatal adverse events | 11 | 10
  Leading to discontinuation of IP | 1 | 3
  Leading to discontinuation from study treatment | 9 | 8

ADVERSE EVENTS:
Time Frame: Approximately 8 weeks (4 treatment cycles)
Description: All participants in the Primary Analysis Set who received at least 1 dose of investigational product were included in the safety analysis set. One participant was randomized to the placebo arm but actually received pegfilgrastim and is included in the pegfilgrastim arm for the safety analyses.
Arm/Group | Placebo | Pegfilgrastim
Serious Adverse Events (participants affected / at risk) | 56/421 | 68/420
Other Adverse Events (participants affected / at risk) | 310/421 | 298/420
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=421) | Pegfilgrastim (N=420)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 5
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 3
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic stenosis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 10
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 4
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Intestinal fistula (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 3
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 3
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 2
Rectal perforation (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 4
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 2 | 0
Hernia (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Medical device complication (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 5
Sudden death (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatorenal failure (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Abscess rupture (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 1 | 1
Device related sepsis (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 1
Kidney infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Oral fungal infection (Infections and infestations) | 1 | 0
Pelvic infection (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 4
Soft tissue infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram abnormal (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Delirium (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 2
Embolism venous (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Phlebitis deep (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=421) | Pegfilgrastim (N=420)
Anaemia (Blood and lymphatic system disorders) | 23 | 34
Neutropenia (Blood and lymphatic system disorders) | 121 | 46
Abdominal pain (Gastrointestinal disorders) | 21 | 25
Constipation (Gastrointestinal disorders) | 47 | 44
Diarrhoea (Gastrointestinal disorders) | 103 | 107
Nausea (Gastrointestinal disorders) | 91 | 115
Stomatitis (Gastrointestinal disorders) | 24 | 9
Vomiting (Gastrointestinal disorders) | 45 | 47
Asthenia (General disorders) | 34 | 31
Fatigue (General disorders) | 64 | 70
Pyrexia (General disorders) | 31 | 56
Weight decreased (Investigations) | 19 | 26
Decreased appetite (Metabolism and nutrition disorders) | 31 | 40
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 23
Neuropathy peripheral (Nervous system disorders) | 25 | 29
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23 | 30
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 25
Hypertension (Vascular disorders) | 28 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.